CLINICAL TRIAL: NCT06606795
Title: The Effects of Cervical and Thoracic Manipulation Therapy Applied to Weightlifting Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Kaan ALTUNOK, Lecturer, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SelcukU_PT_WeightliftingMnp.1
Record Dates: First submitted 2024-09-09; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Weightlifting; Breathing; Breath Tests; Athlete; Spinal Manipulation
Keywords: Weightlifting; Chiropractic; Breathing; Spinal Manipulation; Athlete
MeSH Terms: conditions — Respiratory Aspiration | interventions — Manipulation, Spinal; Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: Individuals will be randomly assigned to control and spinal manipulation groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): 20 people will be included in the control group. A total of two measurements will be taken, one at the beginning and one at the end of the study. Respiratory muscle strength, respiratory function, and cervical and thoracic joint range of motion will be evaluated in the measurements. The control group will continue their normal weightlifting training throughout the study.
- Spinal Manipulation Group (Experimental): 20 people will be included in the Spinal Manipulation Therapy (SMT) group. This group will continue their normal weightlifting training during the study and in addition to the weightlifting training, they will receive a total of three sessions of cervical and thoracic manipulation therapy once a week for three weeks. A total of two measurements will be taken at the beginning and end of the study. Respiratory muscle strength, respiratory function and cervical and thoracic joint range of motion will be evaluated in the measurements.
  Interventions: Other: Spinal Manipulation

INTERVENTIONS:
Other: Spinal Manipulation — For the treatment to be applied in the SMT group, segmental dysfunctions will be determined using static and dynamic palpation techniques and the applications will be applied with a chiropractic method, high-speed, low-amplitude spinal manipulation method, at the level of the dysfunctional spine.
  Other Names: Chiropractic Manipulation
  Arms: Spinal Manipulation Group

SUMMARY:
The effects of manipulation therapy on the autonomic nervous system have been examined in the literature and while no sympathetic or parasympathetic changes were found after upper thoracic manipulation, a decrease in sympathetic data was observed after lower thoracic manipulation and an increase in parasympathetic data was observed. On the other hand, a different study found that thoracic manipulation did not cause any changes such as an increase or decrease in the autonomic nervous system. Therefore, although there are uncertainties in the autonomic role of manipulation therapy, its effect on respiration is intriguing when positive studies are considered.

In a study aiming to evaluate the effect of thoracic manipulation on respiratory function, segmental manipulation treatment was applied to healthy individuals by detecting the vertebrae in the thoracic region where normal joint movements were lost, and it was determined that the respiratory functions of the manipulation group improved significantly compared to the group that did not receive treatment. In another study conducted on healthy individuals, the subjects were divided into manipulation group, exercise and manipulation group and control groups. At the end of the study, it was determined that there was a significant increase in the respiratory functions of the participants in the manipulation group, while an additional increase was observed in the group combined with exercise, but this was not significant. No change was observed in the control group.

When the literature is examined, it is noteworthy that the effects of manipulation treatments on respiration remain unclear, and especially the inadequacy of studies on Olympic-style weightlifters and the ongoing search for increasing athletic performance in this area.

This study aims to examine the effects of cervical and thoracic manipulation treatments on respiratory muscle strength, respiratory functions and cervical and thoracic region joint range of motion in weightlifters.

The main question it aims to answer is:

- Is cervical and thoracic manipulation therapy applied to Olympic style weightlifters effective on respiration?

DETAILED DESCRIPTION:
Our study is planned as a prospective, randomized controlled, single-blind experimental study. A total of 40 female and male elite and non-elite weightlifters between the ages of 13-35 will be evaluated for our study.

The minimum sample size of the study was found to be at least 40 people, with at least 20 people in each group, with 90% power at a 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Being a weightlifter,
* Having asymptomatic dysfunction in the cervical and thoracic spine,
* Not having received any manipulative treatment in the last six months,
* Individuals who do not have a condition that prevents chiropractic manipulation treatment will be included in the study.

Exclusion Criteria:

* Having had an injury related to the musculoskeletal system in the upper and lower extremities in the last month,
* Having any neurological and psychiatric disorders,
* Having cervical disc herniations,
* Having a disorder related to the cardiac and respiratory systems,
* Having an infectious, rheumatological, metabolic and endocrinological disorder,
* Having dislocation, osteoporosis, ankylosing spondylitis, discopathy, rheumatoid arthritis,
* Taking anticoagulant treatment,
* Individuals who have recently undergone an operation involving the cervical and thoracic regions will not be included in the study.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-04 (Estimated); Primary Completion 2024-10-18 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | 3 weeks
  In our study, the respiratory muscle strength of the participants will be measured and recorded as maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) with the help of a portable device that can measure intraoral pressure electronically, which is a non-invasive method. The nose of the participant who makes maximal expiration in the sitting position will be closed with a valve and the MIP measurement will be completed by asking for maximal inspiration for 1-3 seconds and the measurements will be recorded. The nose of the participant who makes maximal inspiration in the sitting position will be closed with a valve and the MEP measurement will be completed by asking for maximal expiration for 1-3 seconds and the measurements will be recorded. The highest of the three best results among at least five measurements with no more than 10% difference between them will be recorded as the final data.
Respiratory function test | 3 weeks
  Respiratory functions will be assessed with a portable spirometer with the patient in a sitting position according to the criteria determined by the American Thoracic Society and the European Respiratory Society. Spirometry measures multiple parameters during a single test. The test will be repeated three times. Participants will be asked to perform a single forced expiration followed by a single inspiration during normal breathing, and with this single measurement; forced expiratory volume in the first second of the respiratory function test (FEV₁), forced vital capacity (FVC), forced expiratory volume in the first second/forced vital capacity ratio (FEV₁/FVC), peak expiratory flow rate (PEF) and forced expiratory midflow rate (FEF%25-75) and the highest and percentages of the expected vital capacity (VC) values after three consecutive tests will be obtained. These results obtained with a single breathing test will be recorded as the highest and percentages of the expected values.
Range of Motion of Cervical and Thoracic Regions | 3 weeks
  A gravity-dependent inclinometer and Spinal Mouse, which have been proven to be reliable in studies, will be used for measurements. Joint motion of the cervical and thoracic regions will be evaluated with the Lafayette brand Acumar Digital Dual Inclinometer and Spinal Mouse.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sillevis R, Cleland J, Hellman M, Beekhuizen K. Immediate effects of a thoracic spine thrust manipulation on the autonomic nervous system: a randomized clinical trial. J Man Manip Ther. 2010 Dec;18(4):181-90. doi: 10.1179/106698110X12804993427126. PMID 22131791
- [Background] Shin DC, Lee YW. The immediate effects of spinal thoracic manipulation on respiratory functions. J Phys Ther Sci. 2016 Sep;28(9):2547-2549. doi: 10.1589/jpts.28.2547. Epub 2016 Sep 29. PMID 27799691
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Engel RM, Vemulpad S. The effect of combining manual therapy with exercise on the respiratory function of normal individuals: a randomized control trial. J Manipulative Physiol Ther. 2007 Sep;30(7):509-13. doi: 10.1016/j.jmpt.2007.07.006. PMID 17870419